CLINICAL TRIAL: NCT02880527
Title: Study of the Prevalence of Polymyositis and Dermatomyositis in Normandy
Acronym: EPIDEMYOSITIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/007/HP
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Polymyositis; Dermatomyositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with polymyositis / dermatomyositis: recruitment of patients with polymyositis / dermatomyositis will be used:
  1. medical specialists , hospital and liberals who support patients with polymyositis / dermatomyositis ( internists , dermatologists, neurologists, pulmonologists , rheumatologists ) ;
  2. general practitioners
  3. the PMSI data for public and private hospitals ; 4 ) data boxes regional health insurance (primary health insurance fund , MSA Normandy , Social Scheme for Self )
  5) Norman patients, members of an association of patients with polymyositis / dermatomyositis : the French Muscular Dystrophy Association
  Interventions: Other: Patients with polymyositis / dermatomyositis

INTERVENTIONS:
Other: Patients with polymyositis / dermatomyositis — recruitment of patients with polymyositis / dermatomyositis using :
  1. medical specialists , hospital and liberals who support patients with polymyositis / dermatomyositis ( internists , dermatologists, neurologists, pulmonologists , rheumatologists ) ;
  2. general practitioners
  3. the PMSI data for public and private hospitals ; 4 ) data boxes regional health insurance (primary health insurance fund , MSA Normandy , Social Scheme for Self )
  5) Norman patients, members of an association of patients with polymyositis / dermatomyositis : the French Muscular Dystrophy Association

SUMMARY:
Polymyositis and dermatomyositis are characterized by the association to a myopathic syndrome, inflammatory infiltrates in the skeletal muscle. They remain, even today, an important factor of morbidity and mortality in these patients. At present, studies that evaluated the prevalence of polymyositis / dermatomyositis are very few; they were mainly recorded in the United States and Japan, the prevalence of polymyositis / dermatomyositis has been estimated between 3.5 and 21.5 cases / 100 000 (according to the old diagnostic criteria of Bohan and Peter). However, previous works are old and retrospective; above all, they have almost always been performed (90% of cases) from cases reported to the hospital, leading to selection bias and an underestimate of the true prevalence of polymyositis / dermatomyositis in the general population.

Thus, these data lead to achieve this epidemiological study, descriptive, multicenter, based on the population of Normandy.

ELIGIBILITY:
Inclusion Criteria:

* patients with polymyositis / dermatomyositis, meeting the diagnostic criteria for ENMC;
* patient living Normandy ;
* patient has been informed and has given its verbal agreement ;

Exclusion Criteria:

* patients with myositis diagnosed before inclusion (including pathophysiology, clinical phenotype and therapeutic care are different from polymyositis / dermatomyositis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in the Normandy with polymyositis / dermatomyositis
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Confirmed diagnosis of polymyositis / dermatomyositis | approximately 1 month
  recruitment of patients with polymyositis / dermatomyositis

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MARIE, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France